CLINICAL TRIAL: NCT00560989
Title: Shared Genetic Susceptibility in CBD and Sarcoidosis
Brief Title: Identifying Shared Genetic Susceptibility Regions in Chronic Beryllium Disease and Sarcoidosis
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1382; R21HL081766 (NIH); R21HL081766-01A2 (NIH)
Record Dates: First submitted 2007-11-16; First posted 2007-11-20 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Sarcoidosis; Berylliosis
Keywords: Chronic Beryllium Disease; CBD; Beryllium; Genetic; Environmental
MeSH Terms: conditions — Sarcoidosis; Berylliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: CBD cases
- 2: Beryllium-exposed, non-diseased control subjects
- 3: Sarcoidosis cases
- 4: Sarcoidosis control subjects

SUMMARY:
Granulomatous lung diseases are diseases in which inflamed clusters of white cells, known as granulomas, form in lung tissue. Chronic beryllium disease (CBD) and sarcoidosis are two granulomatous diseases that share similar clinical symptoms, physiological changes in the lungs, and immune responses to the disease. Genetic variations may make some people more susceptible to developing CBD or sarcoidosis. This study will identify common genetic regions associated with increased risk of developing the granulomatous diseases CBD and sarcoidosis.

DETAILED DESCRIPTION:
CBD and sarcoidosis are granulomatous lung diseases that are caused by an abnormal immune response. While CBD is known to develop from exposure to the industrial product beryllium, the cause of sarcoidosis remains undetermined. CBD occurs in 2 to 16% of people exposed to beryllium and varies in severity of symptoms. People with sarcoidosis often show very minor symptoms. However, certain variables have been associated with the more severe forms of disease. These variables include black race, onset over the age of 40, involvement of more than three affected organs, and presence of more serious lung disease. When serious symptoms of sarcoidosis occur, clinical and pathological appearances of CBD and sarcoidosis are often hard to distinguish. Symptoms common to both diseases include fever, chest pain, weight loss, night sweats, fatigue, and presence of granulomas on the lungs. The fact that the severity of both diseases varies greatly among those affected points to possible genetic involvement. The genetic basis being analyzed in this study begins with the similar immune responses in the development of both diseases, specifically involving human leukocyte antigen (HLA) gene products. The purpose of this study is to identify common genetic regions associated with increased risk of developing the granulomatous diseases CBD and sarcoidosis.

This study will utilize a novel technique, known as a genome-wide scan. The study will examine previously collected DNA samples from participants in a previous NIH study, A Case Control Etiologic Study of Sarcoidosis (ACCESS), and from participants with CBD recruited at the National Jewish Medical and Research Center. Using the genome scans, researchers will compare genetic regions of people with CBD versus people without CBD who have been exposed to beryllium. The same approach will be used to define genetic regions associated with sarcoidosis. Genome control methods will be used to account for population stratification in both the CBD and sarcoidosis populations. Researchers will compare data between diseased and healthy control groups and between CBD and sarcoidosis groups to identify shared genetic regions relevant to disease development. A second genome scan involving two larger populations of CBD and sarcoidosis cases and controls will be conducted to confirm the association of these regions with both diseases.

ELIGIBILITY:
Inclusion Criteria:

* Has previously participated in beryllium studies conducted by Dr. Lisa Maier
* Agrees to allow the use of personal medical records and genetic material for future research by study officials

Exclusion Criteria:

* Will not consent for use of DNA for research purposes or for storage
* Any beryllium or sarcoidosis DNA specimens without an optical density of 260/280 nm, ratio between 1.8 and 2.0, or with an insufficient quantity of DNA for analysis purposes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will use specimens from two well-established disease popultions: a CBD population previously recruited at the National Jewish Medical and Research Center and a sarcoidosis population derived from the previous NHLBI study, A Case-Control Etiologic Study of Sarcoidosis (ACCESS).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2007-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Shared genetic regions associated with the risk of the granulomatous diseases CBD and sarcoidosis | Measured at completion of genetic analysis

SECONDARY OUTCOMES:
Genetic/chromosomal regions associated with CBD and sarcoidosis | Measured at completion of genetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Maier, MD, MSPH, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States